CLINICAL TRIAL: NCT05919485
Title: The Effects of Specific Transcranial Direct Current Stimulation tDCS on Cognition in Mild Cognitive Impairment: A Novel Study Protocol
Brief Title: The Effects of Specific tDCS on Cognition in MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Prof. Dr. MD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023IMU_ALKU
Record Dates: First submitted 2023-06-08; First posted 2023-06-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Parkinson Disease
Keywords: Mild cognitive impairment; Alzheimer's disease; Parkinson's disease; Transcranial direct current stimulation
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The distribution of the sham or real stimulators will be based on the random allocation which makes it impossible to identify the sham or real stimulation for the participants and the test instructors. This double-blind masking procedure will be applied all throughout the study steps in line with the reference study. The randomization data will be confidential and will not be accessible except for the medical emergencies. After the above-mentioned blinding process has been ended, the participants will be managed as off-study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interventional-DLPFC (Experimental): DLPC/F3-F4 group will consist of 20 PD-MCI patients and 20 aMCI patients; 2mA anodal tDCS over DLPFC The current density will be 0.06mA/cm2 from each electrode with total density of 0.054/cm2 and will be delivered for 20 minutes for the atDCS group for 5 days a week, for 10 days and a total of 10 sessions in 14 days.
  Interventions: Procedure: tDCS
- Interventional-LPC (Experimental): LPC/P3-P4 group will consist of 20 PD-MCI patients and 20 aMCI patients; 2mA anodal tDCS over LPC The current density will be 0.06mA/cm2 from each electrode with total density of 0.054/cm2 and will be delivered for 20 minutes for the atDCS group for 5 days a week, for 10 days and a total of 10 sessions in 14 days.
  Interventions: Procedure: tDCS
- Sham (Sham Comparator): Sham control group will consist of 40 patients (20 aMCI and 20 PD-MCI patients).
  2mA anodal sham tDCS protocol. For the sham protocol, the stimulation will be delivered for one time with a very low current frequency, enough to cause slight tingling, and for 15 seconds long which will also be delivered for 20 minutes, 5 days a week, for 10 days and a total of 10 sessions in 14 days.
  Interventions: Procedure: tDCS

INTERVENTIONS:
Procedure: tDCS — 0.06mA/cm2 from each electrode with total density of 0.054/cm2 for 20 minutes for 5 days a week, for 10 days and a total of 10 sessions in 14 days.
  Brain area; DLPFC / LPC

SUMMARY:
INTRODUCTION:

Mild cognitive impairment (MCI) is a critical transitional stage in dementia related disorders. Dorsolateral prefrontal cortex (DLPFC), and the lateral parietal (LPC) cortex are subjected to neuropathological changes in MCI. Parietal memory network (PMN) integrity alterations and default mode network (DMN) alterations also occur in MCI. Transcranial direct current stimulation (tDCS) is a promising neuroprotective tool that modulates functional connectivity and might be useful to interfere with cognitive decline in relation to amnestic MCI (aMCI) and Parkinson's disease-MCI (PD-MCI) when applied to DLPFC and LPC.

METHODS:

This is a multicenter, randomized, and controlled study evaluating the effectiveness of anodal tDCS (atDCS ) applied bilaterally to the DLPFC/F3-F4 and LPC/ P3-P4 for 5 sessions with a total of 10 sessions in 14 days. The stimulation will be delivered with a 2 mA current frequency and will last 20 minutes a day for 5 days a week. The study consists of anodal, and sham control groups with a total of 120 participants with DLPFC and LPC anodal groups including 40 participants each and sham including 40 participants which are all between 45-80 years of age.

At baseline and as an outcome measure, neurocognitive evaluation will be conducted using various tests standardized to use in the Turkish population. Functional magnetic resonance (fMRI) will be used to detect possible PMN and DMN alterations and hippocampal connectivity, and electroencephalogram (EEG) will be used to assess possible electrophysiological alterations that may happen as a result of atDCS. Baseline evaluation will be done before atDCS sessions and it will be repeated at the end of 14 days and 90 days.

DISCUSSION:

This study aims to explore the effectiveness of atDCS in PD-MCI, aMCI and to contribute to the literature in the field.

DETAILED DESCRIPTION:
Study Design This is a multi-center, randomized, controlled study registered and carried out at Medipol University Hospital and Alaaddin Keykubat University Training and Research Hospital. The objective of the study is to evaluate the effectiveness of atDCS stimulation over DLPFC and LPC on cognitive skills of patients with PD-MCI and aMCI.

The patients will be randomized to 2mA tDCS over DLPFC and over LPC, or Sham control. tDCS stimulation will last for 20 minutes a day for 5 consecutive days, a total of 10 sessions in 14 days. The outcome of the simulations will be evaluated by various neurocognitive tests at the baseline, at the end of 14 days and then, 90 days.

Brain connectivity will be analyzed by resting state-functional magnetic resonance imaging (fMRI) and neuronal activity will be analyzed by electroencephalography (EEG) at the baseline, at the end of 14 days and 90 days..

This study aims to give important translational messages in the field of clinical neuroscience by exploring the pro-cognitive effects of tDCS application including its optimal application methods. In this framework, the restorative benefits of tDCS can be critical to understand the cause-effect relationship between certain neural circuits and behavioral outcomes, which might be important in understanding the pathophysiology of MCI and PD. From another point of view, our findings might be valuable in terms of prolonged life-expectancy and the maintenance of preserved cognitive skills in the elderly.

Although tDCS is still in a premature stage, it has certain advantages in terms of portability, cost-effectiveness and user-friendly application compared to other non- invasive stimulation applications. This study will contribute to the growing literature in terms of its optimal application methods, side-effects and long-term (90 days) neurobehavioral results.

ELIGIBILITY:
Inclusion Criteria:

1. Providing an informed consent;
2. Literate and between 45-80 years of age;
3. 60 females and 60 males;
4. Diagnosed with PD based on criteria suggested by UK Parkinson's Disease Society, Brain Bank and PD-MCI in accordance with the diagnostic criteria suggestions by Litvan;
5. Diagnosed with aMCI based on diagnosis criteria (CDR>0.5) suggested by Petersen;
6. On a stable pharmacological treatment minimum for one month with no washout period.

Exclusion Criteria:

* Illiterate or education level less than primary school
* Having an existing and/or prior neurological disease; psychiatric disease or head trauma; and/or irreversible hearing or sight problems or other medical illness (e.g. diabetes mellitus, hypertension);
* Exhibiting signs of dementia for PD group ;
* Having medical issues that prevent undergoing fMRI or for tDCS application.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Tests Scores | Changes Before Treatment and 14 Days&90 Days after treatment
  Moca, AdCom Scores

SECONDARY OUTCOMES:
EEG Power Spectrum Analysis | Changes Before Treatment and 14 Days after treatment
  EEG data will be separated into one-second epochs after they are cleared of noise. Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform (FFT, Fast Fourier Transform) with 10% Hanning window, then power spectrum analysis will be performed, giving the frequency values for each electrode by averaging all FFTs. Maximum peaks will be determined in the delta (0.5-3.5 Hz), theta (4-7 Hz), alpha (8-13 Hz), beta (15-28 Hz) and gamma (28-48 Hz) frequency bands. these values will be used in statistical analysis for each person and electrode.
EEG Coherence Analysis | Changes Before Treatment and 14 Days after treatment
  Coherence measurements at delta, theta, alpha, beta and gamma frequencies can be analyzed for either intra-hemispheric electrode connections or inter-hemipheric electrode connections.Coherence values take values between 0-1. Values close to 0 indicate that there is no connection at the determined frequency between the two calculated electrode regions, while values close to 1 indicate a high coupling between the two electrode regions. Coherence values will be calculated with the Brain Vision Analyzer program using the formula below.The data obtained during memory and visualization will be separated into one-second epochs after they are cleared of noise.Power spectrums of these data will be obtained in the delta, theta, alpha, beta and gamma frequency bands. Each epoch will be analyzed by Fast Fourier Transform with 10% Hanning window.Then, these data will be calculated for all possible electrode pairs using the brain vision analysis program with the formula given below.
EEG functional connectivity analysis | Changes Before Treatment and 14 Days after treatment
  eLORETA software will be used for functional connectivity analysis. sLORETA /eLORETA is an online free software developed by Roberto Pascual-Marqui and his team (http://www.uzh.ch/keyinst/loreta.htm). eLORETA is an algorithm developed to solve the inverse problem and it does not contain localization bias even in the presence of noise . In this software, resting state data with eyes closed, separated into 2 second epochs, whose artifacts are cleaned by preprocessing, will be used. The relevant areas to be analyzed in the cortical plane and the relevant frequency band gaps will be determined. The time series containing the eLORETA current source density obtained from these areas will be calculated and a "lagged linear coherence" matrix will be created to be applied in graph theory (Vecchio et al., 2014). "Lagged linear coherence" will give correct physiological connectivity unaffected by volume conduction and low spatial resolution.
Volumetric Magnetic resonance Imaging (MRI) and functional magnetic resonance imaging (rest-fMRI) | Changes Before Treatment and 14 Days after treatment
  The change in central nervous system atrophy and resting state network activity between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaaddin Keykubat Üniversitesi, Antalya, Alanya, Turkey (Türkiye)